CLINICAL TRIAL: NCT05553106
Title: Evaluation of Cognitive Status, Kinesiophobia, Physical Activity Level, and Functional Performance in Coronary Intensive Care
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dilara Saklica, Principal Investigator, Hacettepe University
Other Study IDs: GO 20/299
Record Dates: First submitted 2022-09-19; First posted 2022-09-23 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Heart Diseases
Keywords: intensive care; coronary artery disease; kinesiophobia; physical activity level
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease; Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Patients who are hospitalized in the coronary intensive care unit, who can take simple commands, and whose condition is physiologically stable.

SUMMARY:
The aim of our study is to evaluate cognitive status, kinesiophobia, physical activity level, and functional performance in coronary intensive care.

DETAILED DESCRIPTION:
This study will be performed on patients who are hospitalized in the coronary intensive care unit, who can take simple commands, and whose condition is physiologically stable.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being under surveillance in the coronary intensive care unit

Exclusion Criteria:

* Presence of neurological disease that may affect the cognitive status
* Not being clinically stable
* Not to cooperate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in coronary intensive care unit who can take simple commands and whose condition is physiologically stable
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Functional Performance Assessment | 2 weeks
  Functional status score for the intensive care unit (FSS-ICU) will be used.

SECONDARY OUTCOMES:
Symptom Assessment | 2 weeks
  Cardiac symptom survey will be used.
Cognitive Status Assessment | 2 weeks
  The Montreal Cognitive Assessment (MoCA) will be used
Physical Activity Level | 2 weeks
  Physical activity level will be evaluated using the International Physical Activity Questionnaire - Short Form (IPAQ-SF).
Fear of Movement | 2 weeks
  Fear of movement will be evaluated using the Fear of Activity in Patients with Coronary Artery Disease (Fact-CAD).

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Vardar-Yagli, PhD, Study Director — Hacettepe University; Hikmet Yorgun, PhD, Study Director — Hacettepe University; Ahmet Hakan Ates, PhD, Study Chair — Hacettepe University; Dilara Saklica, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)